CLINICAL TRIAL: NCT02407639
Title: Randomized, Double-blind Trial of CO2 vs. Air Insufflation in Children Undergoing Colonoscopy
Brief Title: Insufflation in Children Undergoing Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Prof. Dr., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CO2vsAIR
Record Dates: First submitted 2015-03-18; First posted 2015-04-03 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Colonoscopy; Children
Keywords: insufflation; abdominal pain
MeSH Terms: conditions — Abdominal Pain | interventions — Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- co2 arm (Active Comparator): insufflation with CO2
  Interventions: Other: CO2
- air arm (Placebo Comparator): insufflation with air
  Interventions: Other: air

INTERVENTIONS:
Other: CO2 — gas
  Arms: co2 arm
Other: air — air
  Arms: air arm

SUMMARY:
Studies in adults have shown that post-procedural abdominal pain is reduced with the use of CO2 instead of air for insufflation during colonoscopy. The aim of our study is to compare post-procedural abdominal pain and girth in children undergoing colonoscopy using CO2 or air for insufflation.

DETAILED DESCRIPTION:
Several prospective studies in adults have confirmed the efficacy and safety of CO2 insufflation in comparison with atmospheric air insufflation during colonoscopy. CO2 insufflation was associated with decreased post-procedural abdominal pain, which likely stems from the fact that, in comparison to air, absorption of CO2 from the colon is much faster due to a much greater water solubility. Animal studies have also shown that CO2 insufflation results in less disturbance of parietal blood flow due to its potential vasodilating effect. Insufflation of colon with CO2 did not prolong the procedure or lengthen the time to reach the terminal ileum and was proven to be safe in both sedated and non-sedated patients . The use of CO2 for colon insufflation could possibly lead to CO2 retention and increased levels in the blood thus interfering with acid-base balance . However, previous studies reported that carbon dioxide insufflation did not cause increased CO2 levels in the blood or end-tidal CO2 (ETCO2) and complication rates were not increased when using CO2. Because of its advantages CO2 insufflation has become a standard of care in adult colonoscopy.

To the best of our knowledge there are so far no published reports comparing CO2 and air insufflation during colonoscopy in children.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy

Exclusion Criteria:

* PM retardation
* postprocedural complications regarding sedation

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
to compare post-procedural abdominal pain in children undergoing colonoscopy using CO2 or air for insufflation. | 24 hours
  NRS-11 pain scale will be used to assess abdominal pain, ranging from "no pain" marked as 0 point to "worst pain ever" marked as 10 points. Children will be asked to score the amount of pain experienced at 2, 4, and 24 hours after the examination.

SECONDARY OUTCOMES:
to compare post-procedural girth in children undergoing colonoscopy using CO2 or air for insufflation. | 4 hours
  Waist circumferences will be measured before the examination and 10 minutes, and, 2 and 4 hours after the examination. Measurements will be made using tape measure at the level of the umbilicus.

CONTACTS AND LOCATIONS:
Overall Officials: Matjaž Homan, PhD MD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Homan M, Mahkovic D, Orel R, Mamula P. Randomized, double-blind trial of CO2 versus air insufflation in children undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):993-7. doi: 10.1016/j.gie.2015.08.073. Epub 2015 Sep 10. PMID 26363332